CLINICAL TRIAL: NCT06517511
Title: Selinexor in Combination With R-CHOP as the First-line Therapy for TP53-mutated DLBCL Patients: a Single-arm, Multicenter, Phase II Clinical Trial (Smart Trial)
Brief Title: Selinexor in Combination With R-CHOP as the First-line Therapy for TP53-mutated DLBCL Patients (Smart Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fudan University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-333-01
Record Dates: First submitted 2024-07-14; First posted 2024-07-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: TP53-mutated diffuse large B-cell lymphoma; Selinexor
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — selinexor; Exportin 1 Protein; R-CHOP protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Selinexor in combination with R-CHOP (Experimental): Patients with TP53-mutated diffuse large B-cell lymphoma will receive selinexor in combination with R-CHOP regimen from the second cycle of R-CHOP (3 weeks per cycle).
  After 8 cycles of induction therapy, if the response is assessed as complete remission (CR), maintenance therapy with selinexor will be conducted.
  Interventions: Drug: Selinexor Oral Tablet [Xpovio]; Drug: R-CHOP Protocol

INTERVENTIONS:
Drug: Selinexor Oral Tablet [Xpovio] — Selinexor (60mg po D1, 8) is added from the second cycle of R-CHOP regimen.
  Other Names: exportin 1 (XPO1) inhibitor
Drug: R-CHOP Protocol — Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone
  Other Names: R-CHOP regimen

SUMMARY:
This is a prospective, single-arm, multi-center, phase II clinical trial to evaluate the efficacy and safety of selinexor in combination with R-CHOP (rituximab, cyclophosphamide, vincristine, doxorubicin, and prednisone) followed by selinexor maintenance for untreated TP53-mutated diffuse large B-cell lymphoma (DLBCL) patients.

DETAILED DESCRIPTION:
The purpose of this phase II clinical trial is to evaluate the efficacy and safety of selinexor in combination with R-CHOP for untreated TP53-mutated DLBCL patients.

The induction phase consisted of 8 cycles of selinexor in combination with R-CHOP. After 8 cycles of induction therapy, if the response is assessed as complete remission (CR), maintenance therapy with selinexor will be conducted.

The primary endpoint is complete response rate.

ELIGIBILITY:
Inclusion Criteria:

* Subjects fully understand and voluntarily participate in this study and sign informed consent.
* Aged ≥18 and ≤80 years, no gender limitation.
* Histologically confirmed DLBCL with TP53 mutations (allowing transformed or concurrent indolent B-cell non-Hodgkin lymphoma)
* No prior systemic anti-lymphoma therapy; prior local radiotherapy alone is permitted.
* There must be at least one measurable or evaluable lesion that meets the evaluation criteria for Lugano 2014 lymphoma.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2.
* Expected survival ≥ 3 months.
* Adequate function of bone marrow, liver, and kidney.

Exclusion Criteria:

* DLBCL with Hodgkin lymphoma, T-cell lymphoma, or other non-B-cell lymphoma; Richter transformation.
* DLBCL with central nervous system invasion.
* The patients had previously received XPO1 inhibitors.
* The patients have contraindications to any drug in the combined treatment.
* Patients with chronic active hepatitis B or active hepatitis C. If the background hepatitis B surface antigen (HBsAg) and/or hepatitis B core Antibody (HBcAb) or hepatitis C Virus (HCV) antibody are positive, the further determination for Hepatitis B Virus (HBV) DNA (no more than 2500 copies /mL or 500 IU/mL) and HCV RNA (no more than the lower limit of the assay) can be included. The patients with HBsAg and/or HBcAb positive need to receive anti-HBV drugs.
* Patients with the infection of human immunodeficiency virus (HIV) and/or acquired immunodeficiency syndrome.
* Inability to swallow tablets, presence of malabsorption syndrome, or any other gastrointestinal disease or dysfunction that may affect the absorption of the study drug.
* Pregnant and lactating women and subjects of childbearing age who do not want to use contraception.
* Mentally ill persons or persons unable to obtain informed consent.
* Any condition deemed unsuitable by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Complete response rate (CRR) | Up to 8 cycles (each cycle is 21 days)
  To investigate the preliminary anti-tumor efficacy

SECONDARY OUTCOMES:
Disease-free survival (DFS) | From date of the first complete response until the date of the first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  To investigate the preliminary anti-tumor efficacy
Objective response rate (ORR) | Up to 8 cycles (each cycle is 21 days)
  To investigate the preliminary anti-tumor efficacy
Progression-free survival (PFS) | From the date of enrollment until the date of the first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  To investigate the preliminary anti-tumor efficacy
Overall survival (OS) | From the date of enrollment until the date of death from ant cause, assessed up to 24 months
  To investigate the preliminary anti-tumor efficacy
Number of participants with adverse events (AE) and severe adverse events (SAE) as assessed by CTCAE v5.0 | Through study completion, an average of 2 years
  To identify the incidence of AE and SAE
Duration of response (DOR) | From date of the first CR or PR to the first documented progressive disease or death, whichever occurred earlier, assessed up to 24 months
  To investigate the preliminary anti-tumor efficacy
Time to response (TTR) | From the date of enrollment until the first response, assessed up to 24 weeks
  To investigate the preliminary anti-tumor efficacy

OTHER OUTCOMES:
The gene mutations such as DDX3X、TET2、PTPN2 and so on are sequenced by whole genome sequencing | Through study completion, an average of 2 years
  To explore the correlations between gene mutations and response and prognosis
The RNA alterations are sequenced by transcriptome sequencing | Through study completion, an average of 2 years
  To explore the correlations between RNA alterations and response and prognosis
Genetic classification of DLBCL | Through study completion, an average of 2 years
  To explore the correlations between genetic classification of DLBCL and response and prognosis

CONTACTS AND LOCATIONS:
Overall Officials: QingQing Cai, MD. PhD., Principal Investigator — Sun yat-sen university cancer cente; Yi Xia, MD. PhD., Principal Investigator — Sun yat-sen university cancer cente; Rong Tao, MD., Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Sun yat-sen university cancer center, Guangzhou, Guangdong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality